CLINICAL TRIAL: NCT03782779
Title: Respiratory Physical Therapy Based on Diaphragmatic Breathing Program In Institutionalized Older People
Brief Title: Diaphragmatic Breathing Program In Older People
Acronym: BP-OP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Anna Arnal, PhD, Profesora Ayudante, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ID001
Record Dates: First submitted 2018-12-14; First posted 2018-12-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Aging
Keywords: Respiratory physical therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing program and regular exercise (Experimental): Diaphragmatic Breathing Program plus regular upper and lower limb exercises
  Interventions: Other: Breathing program and regular exercise
- Regular Exercise (Active Comparator): Regular upper and lower limb exercises
  Interventions: Other: Regular Exercise

INTERVENTIONS:
Other: Breathing program and regular exercise — This program will be supervised by a physical therapist and will include learning and performing a diaphragmatic-abdominal breathing, and incorporating the new breathing pattern to a upper and lower limbs regular exercises as well as to daily life activities.
  Arms: Breathing program and regular exercise
Other: Regular Exercise — Regular upper and lower limbs exercises supervised by a physical therapist
  Arms: Regular Exercise

SUMMARY:
In the present study a program of respiratory physical therapy based on diaphragmatic breathing is applied in institutionalized old people, evaluating lung function parameters (FVC, FEV1, FEV1/FVC) and oxygen saturation.

The hypothesis is that a diaphragmatic breathing program applied in elderly people can improve the respiratory system's function and consequently improve their daily life. This program will include learning and performing a diaphragmatic-abdominal breathing, and incorporating the new breathing pattern to a upper and lower limbs maintenance exercises as well as to daily life activities.

Methods: randomized and controlled clinical study of respiratory parameters of institutionalized old people. The subjects will be divided into 2 groups: 1) diaphragmatic breathing program and upper and lower limbs maintenance exercises 2) control group which do upper and lower limbs maintenance exercises. There will be 3 treatment sessions during 8 weeks, with evaluations before the study and after 8 weeks, which include: lung function parameters (forced vital capacity, forced expiratory volume in one second, Tiffeneau Index) and pulseoximeter (which includes oxygen saturation and cardiac frequency).

DETAILED DESCRIPTION:
Introduction.The aging of the respiratory system includes physiological changes of the lung as well as the osteoarticular and muscular tissues. Therefore, the European and North American Respiratory Societies highlight in their recommendations the importance of prevention of respiratory diseases. They also insist on the need to maintain the integrity of the anatomical elements that participate in the thoraco-abdominal movements and on preventive treatments in those at risk before the symptoms appear.

Objective. The main objective of this study is to apply a program of supervised breathing program in old people with no respiratory health issues and evaluate the effects on respiratory variables such as forced vital capacity (FVC) forced expiratory volume in one second (FEV1) Tiffeneau Index (FEV1/FVC) and oxygen satutarion (SO2).

Material and Methods Sample: over 60 year old subjects, institutionalized and with no respiratory condition.

Study design. Randomized clinical trial with 2 groups: Group 1. diaphragmatic breathing program and upper and lower limbs maintenance exercises ; Group 2. control group which only do upper and lower limbs maintenance exercises.

Evaluations. Clinical interview with anthropometric data and health characteristics.

There will be 2 evaluations: at the beginning of the study and at the end of the supervised program (at 8 weeks).

In addition, it includes the following evaluation instruments:

* Mini-mental State Examination (MMSE)
* Spirometry: obtaining FVC, FEV1, FEV1/FVC.
* Pulse oxymetry: it measure the SaO2 and cardiac frequency.

ELIGIBILITY:
Inclusion Criteria:

* institutionalized subjects older than or equal to 60 years
* without respiratory pathology diagnosed
* with adequate cognitive status to follow the protocol of respiratory exercises (MEC>30) .

Exclusion Criteria:

* subjects with respiratory diseases
* Subjects with musculoskeletal injuries that prevented the performance of the exercise protocol were excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Forced spirometry | 8 weeks
  Assessed using a COSMED PONY FX spirometer with mouthpiece and filters (1 cardboard mouthpiece and a bacteriological filter per patient). The test was performed with the person sitting, without crossing the legs and shoulders relaxed. Anthropometric data were entered into the equipment, nose was covered with a nose clio and the patient was then asked to perform three forced inhalations and exhalations.
Pulse oxymetry | 8 weeks
  To assess oxygen saturation, a SmartOx pulse oximeter (WEINMANN Medical Technology) is used. The subject remains seated, the pulse oximeter clamp placed on a finger of one of the hands, waiting for the SaO2 and CF value to stabilize and register the value.

SECONDARY OUTCOMES:
Minimental State Examination Folstein | first week
  Mini-Cognitive Lobo est (MEC). To assess the cognitive status before inclusion in the study, the spanish version of Folstein's Minimental State Examination is used. Adapted and validated by Lobo in Spain in 1979. It is a brief cognitive test that consists of the evaluation of the most important cognitive areas (orientation, concentration, calculation, memory, language and construction) with a global maximum score of 35 (30-35 = normal, 24-29 = borderline, <24 in people over 65). The MEC has widely shown its reliability, validity and discriminative power, with a specificity of 75.1% and a sensitivity of 89.8%.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Arnal-Gómez, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain